CLINICAL TRIAL: NCT01439347
Title: Phase 3 Study of Study to Evaluate Marqibo® in the Combination Chemotherapy in the Treatment of Subjects >or=60 Years Old With Newly Diagnosed Acute Lymphoblastic Leukemia (ALL)
Brief Title: A Phase 3 Study to Evaluate Marqibo® in the Treatment of Subjects ≥ 60 Years Old With Newly Diagnosed ALL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTX404
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
Keywords: Marqibo; HALLMARQ; leukemia; front-line; ALL; acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vincristine Sulfate Injection (VSI) (Experimental): VSI dosed at 1.4 mg/m^2 with a 2 mg dose cap as an intravenous (IV) infusion over 10 minutes.
  Interventions: Drug: Vincristine Sulfate Injection (VSI)
- Marqibo (Experimental): Marqibo dosed at 2.25 mg/m^2 (without any dose cap) as an IV infusion over 60 minutes.
  Interventions: Drug: Vincristine Sulfate Liposomes Injection (VSLI)

INTERVENTIONS:
Drug: Vincristine Sulfate Liposomes Injection (VSLI) — 2.25 mg/m^2 (without any dose cap) as an IV infusion over 60 minutes.
  Other Names: Marqibo
  Arms: Marqibo
Drug: Vincristine Sulfate Injection (VSI) — 1.4 mg/m^2 with a 2 mg dose cap as an IV infusion over 10 minutes.
  Other Names: Vincristine
  Arms: Vincristine Sulfate Injection (VSI)

SUMMARY:
A phase 3 study in the treatment of subjects >or= 60 years old with newly diagnosed acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
A phase 3, multicenter, randomized study to evaluate the substitution of Marqibo® (Vincristine Sulfate Liposomes Injection, VSLI) for standard Vincristine Sulfate Injection (VSI) in the induction, intensification, and maintenance phases of combination chemotherapy in the treatment of subjects >or= 60 years old with newly diagnosed acute lymphoblastic leukemia (ALL).

ELIGIBILITY:
Inclusion Criteria:

Have provided written, signed, and dated informed consent to participate in the study, in accordance with the International Council on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice (ICH GCP) Guideline E6 and all applicable local regulations. Are age >or=60 years (at the time of providing informed consent).

Have newly diagnosed, histologically proven, untreated Philadelphia chromosome-negative (Ph-) Acute lymphocytic leukemia [ALL], with >or= 5% bone marrow blasts.

Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. Have a life expectancy >or= 3 months.

Have renal and liver function as defined below within 14 days, inclusive, prior to study enrollment, unless the abnormality is considered attributable to leukemia:

Total bilirubin ≤ 2.0 x the upper limit of normal (ULN), unless the subject has a known diagnosis of Gilbert's disease Aspartate transaminase (AST, Serum glutamic oxaloacetic transaminase [SGOT]) or alanine transaminase (ALT, Serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x ULN Serum creatinine ≤ 1.5 x ULN. Not have had major surgery within 4 weeks before the planned start of treatment.

If female, are post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (eg, hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from the screening visit through 30 days after the last dose of any protocol defined chemotherapeutic agents.

If male and sexually active with a partner of child-bearing potential, agree to use an acceptable barrier method for contraception from the screening visit through 30 days after the last dose of any protocol defined chemotherapeutic agents.

Have the ability and willingness to fully comply with study procedures and restrictions.

-

Exclusion Criteria:

Has had prior systemic chemotherapy (for ALL or other malignancy). Has had prior vincristine for any reason. Is planning to undergo stem cell transplantation (SCT) as any part of first-line therapy for ALL.

Has Burkitt's lymphoma/leukemia. Has Philadelphia chromosome-positive (Ph+) ALL and/or BCR/ABL rearrangements documented by fluorescent in-situ hybridization (FISH), cytogenetics, or polymerase chain reaction (PCR).

Has active central nervous system (CNS) disease. Has ongoing neuropathy of any etiology > Grade 1. Has a history of persistent active neurologic disorders including demyelinating form of Charcot-Marie-Tooth syndrome, acquired demyelinating disorders, and other demyelinating conditions.

Prior hydroxyurea (Hydrea®) for the management of any condition other than leukocytosis or prior hydroxyurea of >7 days duration for the management of leukocytosis (hydroxyurea for the management of leukocytosis must be planned to be tapered off before or on Day 5 of Induction).

Has received prior steroids within 7 days before beginning protocol-specified Induction therapy for reasons other than leukocytosis (steroids for the management of leukocytosis are allowed but must be planned to be tapered off before or on Day 5 of Induction).

Has an active serious infection not controlled by oral or IV antibiotics or antifungals.

Has received any investigational therapy within 28 days before beginning any protocol-defined chemotherapeutic treatment.

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M O'Brien, MD, Principal Investigator — MD Anderson
Locations (15):
- United States (15):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA, Los Angeles, California
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University Fienberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cornell, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vincristine Sulfate Injection (VSI) | Marqibo
Started | 13 | 13
Completed | 0 | 0
Not Completed | 13 | 13
Not completed — Death | 10 | 9
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Terminated Study | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vincristine Sulfate Injection (VSI) | Marqibo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 77] | 67 [60 to 75] | 67 [60 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of study randomization until death from any cause. Observations censored at the date of the last follow-up for subjects not known to have died.
Time Frame: 36 months
Population: Data for this outcome measure was not collected due to early termination of study.
Arm/Group | Vincristine Sulfate Injection (VSI) | Marqibo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Vincristine Sulfate Injection (VSI): VSI dosed at 1.4 mg/m^2 with a 2 mg dose cap as an IV infusion over 10 minutes.
Arm/Group | Vincristine Sulfate Injection (VSI) | Marqibo
All-Cause Mortality (participants affected / at risk) | 10/13 | 9/13
Serious Adverse Events (participants affected / at risk) | 8/13 | 12/13
Other Adverse Events (participants affected / at risk) | 12/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vincristine Sulfate Injection (VSI) (N=13) | Marqibo (N=13)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Sepsis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 1 | 3
Septic Shock (Infections and infestations) | 2 | 2
Bacteraemia (Infections and infestations) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Hepatic Failure (Hepatobiliary disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Blood Bilirubin Increased (Investigations) | 2 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1
Bronchial Secretion Retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Aspergillus Infection (Infections and infestations) | 1 | 0
Cellulitis Orbital (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Transaminases Increased (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vincristine Sulfate Injection (VSI) (N=13) | Marqibo (N=13)
Anaemia (Blood and lymphatic system disorders) | 9 | 6
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 7
Neutropenia (Blood and lymphatic system disorders) | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 9
Constipation (Gastrointestinal disorders) | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 5
Nausea (Gastrointestinal disorders) | 8 | 10
Vomiting (Gastrointestinal disorders) | 5 | 7
Asthenia (General disorders) | 4 | 7
Fatigue (General disorders) | 7 | 3
Oedema Peripheral (General disorders) | 3 | 9
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 6
Alanine Aminotransferase Increased (Investigations) | 5 | 7
Aspartate Aminotransferase Increased (Investigations) | 5 | 7
Blood Alkaline Phosphatase Increased (Investigations) | 5 | 5
Blood Bilirubin Increased (Investigations) | 3 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 7
Hypokalelmia (Metabolism and nutrition disorders) | 6 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 6
Headache (Nervous system disorders) | 6 | 5
Anxiety (Psychiatric disorders) | 5 | 5
Insomnia (Psychiatric disorders) | 4 | 6
Hypotension (Vascular disorders) | 5 | 7
Abdominal Pain (Gastrointestinal disorders) | 4 | 3
Mucosal Inflammation (General disorders) | 3 | 5
Pyrexia (General disorders) | 3 | 3
Lipase Increased (Investigations) | 4 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 3 | 6
Neuropathy Peripheral (Nervous system disorders) | 4 | 4
Paraesthesia (Nervous system disorders) | 4 | 2
Confusional State (Psychiatric disorders) | 2 | 4
Renal Injury (Renal and urinary disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Coagulopathy (Blood and lymphatic system disorders) | 0 | 3
Atrial Fibrillation (Cardiac disorders) | 2 | 2
Palpitations (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Vision Blurred (Eye disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Flatulence (Gastrointestinal disorders) | 1 | 2
Abdominal Distension (Gastrointestinal disorders) | 3 | 1
Chest Pain (General disorders) | 1 | 3
Chills (General disorders) | 3 | 2
Gait Disturbance (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 3
Oedema (General disorders) | 2 | 3
Candida Infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 2
Oral Candidiasis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Blood Creatinine Increased (Investigations) | 0 | 5
Transaminases Increased (Investigations) | 1 | 3
White Blood Cell Count Decreased (Investigations) | 2 | 3
Blood Phosphorus Increased (Investigations) | 3 | 1
Weight Decreased (Investigations) | 2 | 1
Alkaline Phosphatase Increased (Investigations) | 0 | 2
Amylase Increased (Investigations) | 3 | 1
Blood Fibrinogen Decreased (Investigations) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 2 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 1
Neuralgia (Nervous system disorders) | 0 | 2
Neuropathy (Nervous system disorders) | 0 | 3
Syncope (Nervous system disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 2
Mental Status Changes (Psychiatric disorders) | 2 | 3
Agitation (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2
Orthostatic Hypotension (Vascular disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 3 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 1
Bacteraemia (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 1
Chest Discomfort (General disorders) | 2 | 1
Generalised Oedema (General disorders) | 2 | 1
Pain (General disorders) | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1
Oral Pain (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Hepatic Encephalopathy (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No